CLINICAL TRIAL: NCT01959633
Title: Phase I-II Study of the Combination Vemurafenib Plus Cobimetinib Plus PEG-interferon in Advanced Melanoma Patients Harboring the V600BRAF Mutation
Brief Title: Vemurafenib Plus Cobimetinib Plus PEG-interferon in Advanced Melanoma Patients Harboring the V600BRAF Mutation
Acronym: VEMUPLINT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Melanoma Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEMUPLINT; 2013-003730-33 (EudraCT Number)
Record Dates: First submitted 2013-09-27; First posted 2013-10-10 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2019-06

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vemurafenib+Cobimetinib + Peg-interferon (Experimental): Vemurafenib 960 mg b.i.d. + Cobimetinib 60 mg o.d.(21 days on followed by 7 days off) + Peg-interferon 1/2/3 micrograms/Kg once weekly
  Interventions: Drug: Vemurafenib; Drug: Peg-interferon; Drug: Cobimetinib

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib 960 mg b.i.d. for each course of treatment lasting 28 days
  Other Names: Brand name= Zelboraf
Drug: Peg-interferon — In the Phase I are included 3 cohorts. Cohort 1) Peg-interferon 1 µg/Kg one time per week s.c. Cohort 2) Peg-interferon 2 µg/Kg one time per week s.c. Cohort 3) Peg-interferon 3 µg/Kg one time per week s.c. Interferon treatment should start after 15 days of Vemurafenib only
  In the Phase II is included the cohort selected by phase I due to MTD and expanded at RD.
  Other Names: Brand name= Sylatron
Drug: Cobimetinib — Cobimetinib 60 mg o.d. (21 days on followed by 7 days off)
  Other Names: Brand name=Cotellic

SUMMARY:
The hypothesis of this study is to evaluate the safety and the efficacy of Vemurafenib/PEG-interferon combination and the IFNAR1 upregulation lead by this treatment.

DETAILED DESCRIPTION:
Phase I A cohort of 3 consecutive patients will be treated at each dose level (first step). Patients are scheduled to receive at least two courses of therapy (cycle every 28 days) at the same dose level. Escalation of the dose to the next higher level proceeds in absence of dose-limiting toxicity (DLT). Drug-related toxicities will be evaluated during each cycle of therapy and graded according to the NCI Common Toxicity Criteria.

Adverse events (AEs) and the activity of the treatment in terms of ORR, will be assessed as primary endpoints, respectively for phase I and phase II; other variables will be compared as secondary endpoints.

The treatment scheme is Peg-Interferon 1/2/3 micrograms/Kg (lyophilized powder 296 and 444 μg vials) one time per week + Vemurafenib film-coated capsules 960 mg b.i.d. + Cobimetinib tablets 60 mg o.d. 21 days on followed by 7 days off.

Interferon treatment should start after 15 days of Vemurafenib + Cobimetinib only.

Phase I will be conducted at Istituto Nazionale per lo Studio e la Cura dei Tumori - Fondazione G. Pascale (PI Paolo Antonio Ascierto) and a minimum of 3 patients per cohort will be enrolled. Groups of 3 patients will be entered at each dose level (vemurafenib 960 mg b.i.d. + Cobimetinib 60 mg o.d. 21 days on followed by 7 days off + Peg-interferon 1/2/3 micrograms/Kg). DLT will be determined after 2 courses of therapy: if all 3 patients treated at a dose level have been observed for 2 courses of therapy without DLT, then the dose will be escalated. If at least 2/3 patients have DLT after the first 2 courses of therapy in each cohort, then the previous dose level will be considered as the MTD. If 1/3 patients have DLT, then 3 more patients will be treated at this dose level. If none of these patients has DLT, then the dose will be escalated. If at least one of the 3 additional patients has DLT, then the previous dose will be considered the MTD.

The maximum tolerated dose (MTD) is then considered the recommended dose for further evaluation (next step).

Patients experiencing toxicities that were not dose-limiting can be retreated at the same dose level upon full recovery.

Special case is represented by patients with liver metastases for whom ALT or AST increases >3xULN (i.e., Grade 2 of the CTCAE) requires a closer monitoring of the liver tests. In such cases patients with AT up to 5xULN may be allowed to participate in the trial. Therefore, a threshold level of ALT or AST >3xBaseline value (vs. the standard >3xULN threshold) is considered to prompt closer monitoring for the whole duration of the treatment. Patients with rapidly rising or high serum ALT or AST or with ALT or AST elevations accompanied by jaundice require urgent evaluation to find treatable causes of hepatocellular necrosis.

Patients will be treated until progression if the MTD is not reached.

Phase II Phase II will be conducted in approximately 10 Investigational sites located in Italy and 42 patients will be enrolled in total (including 3 patients from the phase I).

Treatment will be continued until progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18
2. Untreated and pretreated (no more than 1 treatment) patients with metastatic melanoma at stage unreseactable IIIb-IV, histologically confirmed, that show V600 type BRAF mutations. Patients eligible for Phase I may have been pretreated with the investigational study treatments.
3. Patient with measurable disease by RECIST v 1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 - 1
5. Patients who have successfully completed all the secondary side effects to previous systemic therapy
6. Patients with an appropriate hematologic, hepatic and renal functionality, assessed in the 7 days preceding the start of therapy, as well as:

   * Absolute neutrophil count (ANC)> 1.5 X 109 / L
   * Absolute platelet count > 100 X 109 / L
   * Hemoglobin > 9 g/dl
   * Serum creatinine < 1.5 times the normal maximum values or Creatinine Clearance > 50 mL/hr (Cockroft-Gault formula)
   * Transaminase level (AST and ALT) < 2.5 times the normal maximum values
   * Serum bilirubin < 1.5 times the normal maximum values
7. Negative pregnancy test performed within 7 days before beginning therapy (premenopausal women)
8. Patients of childbearing age (or with partners of childbearing age) must use effective contraception during therapy and for at least 6 months after the effective treatment
9. Absence of any psychological, familiar or social condition that may affect compliance with study protocol and scheduled follow-up
10. Dated and signed informed consent before any study procedure

Exclusion Criteria:

1. Presence of symptomatic brain metastases
2. Previous malignant cancer during the 2 years preceding the signing of informed consent
3. Investigational study treatment within 28 days or 5 half-lives, whichever is longer, preceding the first dose of study treatments in this study
4. Pregnancy and/or breast feeding;
5. Nausea and vomit refractory to therapy, malabsorption, external biliary shunt, previous bowel resection, which could impair an adequate absorption
6. Any of these conditions occurring in the 6 months before the start of Vemurafenib therapy: heart attack, unstable angina and/or severe degree, congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, arterial hypertension not adequately controlled
7. History of atrial or ventricular arrhythmia, symptomatic> grade 2 (NCI CTCAE)
8. Hystory of retinopathy
9. Correct QT interval > 450msec to baseline history of congenital long QT syndrome
10. Uncontrolled medical condition among which endocrine disorders (such as hypothyroidism, hyperthyroidism and diabetes mellitus)
11. Other severe medical or psychiatric conditions or abnormalities of laboratory tests that may increase the risk associated with study participation or the assumption of Vemurafenib, or that may interfere with the interpretation of study results, which in the judgment of the Investigator can make the patient not eligible for the study
12. Unwillingness to practice adequate contraception
13. Prior systemic treatment with BRAFi or MEKi, or interferon alpha

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | up to 24 weeks
  The NCI CTC-AE (Version 4) will be used to evaluate the clinical safety of the treatment in this study. Patients will be assessed for AEs at each clinical visit up to 24 weeks and as necessary throughout the study.
  Hematology and biochemistry will be done as part of regular safety assessments

SECONDARY OUTCOMES:
Number of Objective tumor responses | From date of randomization until the date of first documented progression or date of death for many cause, whichever came first, assessed up to week 32
  Objective tumor response will be measured according to the modified RECIST 1.1 criteria. Response criteria are essentially based on a set of measurable lesions identified at baseline as target lesions, and followed until disease progression. Durable response rate (DRR) will be identified as the percentage of patients that is still in CR and PR at week 32. The results will be tabulated with Clopper-Pearson 95%CI for response rates

CONTACTS AND LOCATIONS:
Overall Officials: Paolo A Ascierto, MD, Study Chair — Fondazione Melanoma Onlus
Locations (1):
- Fondazione G.Pascale, Napoli, Italy

REFERENCES:
- [Background] Bukowski RM, Tendler C, Cutler D, Rose E, Laughlin MM, Statkevich P. Treating cancer with PEG Intron: pharmacokinetic profile and dosing guidelines for an improved interferon-alpha-2b formulation. Cancer. 2002 Jul 15;95(2):389-96. doi: 10.1002/cncr.10663. PMID 12124839
- [Background] Eggermont AM, Suciu S, MacKie R, Ruka W, Testori A, Kruit W, Punt CJ, Delauney M, Sales F, Groenewegen G, Ruiter DJ, Jagiello I, Stoitchkov K, Keilholz U, Lienard D; EORTC Melanoma Group. Post-surgery adjuvant therapy with intermediate doses of interferon alfa 2b versus observation in patients with stage IIb/III melanoma (EORTC 18952): randomised controlled trial. Lancet. 2005 Oct 1;366(9492):1189-96. doi: 10.1016/S0140-6736(05)67482-X. PMID 16198768
- [Background] Eggermont AM, Suciu S, Santinami M, Testori A, Kruit WH, Marsden J, Punt CJ, Sales F, Gore M, MacKie R, Kusic Z, Dummer R, Hauschild A, Musat E, Spatz A, Keilholz U; EORTC Melanoma Group. Adjuvant therapy with pegylated interferon alfa-2b versus observation alone in resected stage III melanoma: final results of EORTC 18991, a randomised phase III trial. Lancet. 2008 Jul 12;372(9633):117-126. doi: 10.1016/S0140-6736(08)61033-8. PMID 18620949
- [Background] Eggermont AM, Suciu S, Testori A, Santinami M, Kruit WH, Marsden J, Punt CJ, Sales F, Dummer R, Robert C, Schadendorf D, Patel PM, de Schaetzen G, Spatz A, Keilholz U. Long-term results of the randomized phase III trial EORTC 18991 of adjuvant therapy with pegylated interferon alfa-2b versus observation in resected stage III melanoma. J Clin Oncol. 2012 Nov 1;30(31):3810-8. doi: 10.1200/JCO.2011.41.3799. Epub 2012 Sep 24. PMID 23008300
- [Background] Glue P, Fang JW, Rouzier-Panis R, Raffanel C, Sabo R, Gupta SK, Salfi M, Jacobs S. Pegylated interferon-alpha2b: pharmacokinetics, pharmacodynamics, safety, and preliminary efficacy data. Hepatitis C Intervention Therapy Group. Clin Pharmacol Ther. 2000 Nov;68(5):556-67. doi: 10.1067/mcp.2000.110973. PMID 11103758
- [Background] Hwu WJ, Panageas KS, Menell JH, Lamb LA, Aird S, Krown SE, Williams LJ, Chapman PB, Livingston PO, Wolchok JD, Houghton AN. Phase II study of temozolomide plus pegylated interferon-alpha-2b for metastatic melanoma. Cancer. 2006 Jun 1;106(11):2445-51. doi: 10.1002/cncr.21909. PMID 16639739
- [Background] Helfrich I, Edler L, Sucker A, Thomas M, Christian S, Schadendorf D, Augustin HG. Angiopoietin-2 levels are associated with disease progression in metastatic malignant melanoma. Clin Cancer Res. 2009 Feb 15;15(4):1384-92. doi: 10.1158/1078-0432.CCR-08-1615. PMID 19228739
- [Background] Sumimoto H, Hirata K, Yamagata S, Miyoshi H, Miyagishi M, Taira K, Kawakami Y. Effective inhibition of cell growth and invasion of melanoma by combined suppression of BRAF (V599E) and Skp2 with lentiviral RNAi. Int J Cancer. 2006 Jan 15;118(2):472-6. doi: 10.1002/ijc.21286. PMID 16052531
- [Background] Artale S, Sartore-Bianchi A, Veronese SM, Gambi V, Sarnataro CS, Gambacorta M, Lauricella C, Siena S. Mutations of KRAS and BRAF in primary and matched metastatic sites of colorectal cancer. J Clin Oncol. 2008 Sep 1;26(25):4217-9. doi: 10.1200/JCO.2008.18.7286. No abstract available. PMID 18757341
- [Background] Leyton J, Smith G, Lees M, Perumal M, Nguyen QD, Aigbirhio FI, Golovko O, He Q, Workman P, Aboagye EO. Noninvasive imaging of cell proliferation following mitogenic extracellular kinase inhibition by PD0325901. Mol Cancer Ther. 2008 Sep;7(9):3112-21. doi: 10.1158/1535-7163.MCT-08-0264. PMID 18790789
- [Background] Forbes SA, Tang G, Bindal N, Bamford S, Dawson E, Cole C, Kok CY, Jia M, Ewing R, Menzies A, Teague JW, Stratton MR, Futreal PA. COSMIC (the Catalogue of Somatic Mutations in Cancer): a resource to investigate acquired mutations in human cancer. Nucleic Acids Res. 2010 Jan;38(Database issue):D652-7. doi: 10.1093/nar/gkp995. Epub 2009 Nov 11. PMID 19906727
- [Background] Rubinstein JC, Sznol M, Pavlick AC, Ariyan S, Cheng E, Bacchiocchi A, Kluger HM, Narayan D, Halaban R. Incidence of the V600K mutation among melanoma patients with BRAF mutations, and potential therapeutic response to the specific BRAF inhibitor PLX4032. J Transl Med. 2010 Jul 14;8:67. doi: 10.1186/1479-5876-8-67. PMID 20630094
- [Background] Bollag G, Hirth P, Tsai J, Zhang J, Ibrahim PN, Cho H, Spevak W, Zhang C, Zhang Y, Habets G, Burton EA, Wong B, Tsang G, West BL, Powell B, Shellooe R, Marimuthu A, Nguyen H, Zhang KY, Artis DR, Schlessinger J, Su F, Higgins B, Iyer R, D'Andrea K, Koehler A, Stumm M, Lin PS, Lee RJ, Grippo J, Puzanov I, Kim KB, Ribas A, McArthur GA, Sosman JA, Chapman PB, Flaherty KT, Xu X, Nathanson KL, Nolop K. Clinical efficacy of a RAF inhibitor needs broad target blockade in BRAF-mutant melanoma. Nature. 2010 Sep 30;467(7315):596-9. doi: 10.1038/nature09454. PMID 20823850
- [Background] Yang H, Higgins B, Kolinsky K, Packman K, Go Z, Iyer R, Kolis S, Zhao S, Lee R, Grippo JF, Schostack K, Simcox ME, Heimbrook D, Bollag G, Su F. RG7204 (PLX4032), a selective BRAFV600E inhibitor, displays potent antitumor activity in preclinical melanoma models. Cancer Res. 2010 Jul 1;70(13):5518-27. doi: 10.1158/0008-5472.CAN-10-0646. Epub 2010 Jun 15. PMID 20551065
- [Background] Flaherty KT, Puzanov I, Kim KB, Ribas A, McArthur GA, Sosman JA, O'Dwyer PJ, Lee RJ, Grippo JF, Nolop K, Chapman PB. Inhibition of mutated, activated BRAF in metastatic melanoma. N Engl J Med. 2010 Aug 26;363(9):809-19. doi: 10.1056/NEJMoa1002011. PMID 20818844
- [Derived] Simeone E, Scognamiglio G, Capone M, Giannarelli D, Grimaldi AM, Mallardo D, Madonna G, Curvietto M, Esposito A, Sandomenico F, Sabbatino F, Bayless NL, Warren S, Ong S, Botti G, Flaherty KT, Ferrone S, Ascierto PA. A monocentric phase I study of vemurafenib plus cobimetinib plus PEG-interferon (VEMUPLINT) in advanced melanoma patients harboring the V600BRAF mutation. J Transl Med. 2021 Jan 6;19(1):17. doi: 10.1186/s12967-020-02680-7. PMID 33407577